CLINICAL TRIAL: NCT02972177
Title: Clinical Study of Navigation Bronchoscopy Guided Ablation for the Treatment of Peripheral Lung Tumor
Brief Title: Transbronchial Ablation for Peripheral Lung Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE201603
Record Dates: First submitted 2016-11-12; First posted 2016-11-23 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Transbronchial ablation; Radiofrequency ablation; Microwave ablation
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation group (Experimental): Patients with inoperable peripheral lung tumor will be performed transbronchial radiofrequency ablation with the guidance of navigation bronchoscopy. Post treatment response will be evaluated and follow up will be carried out according to the standard procedure.
  Interventions: Procedure: Radiofrequency ablation
- Microwave ablation group (Experimental): Patients with inoperable peripheral lung tumor will be performed transbronchial microwave ablation with the guidance of navigation bronchoscopy. Post treatment response will be evaluated and follow up will be carried out according to the standard procedure.
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Transbronchial radiofrequency ablation will be performed under the guidance of navigation bronchoscopy.
  Arms: Radiofrequency ablation group
Procedure: Microwave ablation — Transbronchial microwave ablation will be performed under the guidance of navigation bronchoscopy.
  Arms: Microwave ablation group

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of navigation bronchoscopy guided transbronchial ablation for the treatment of inoperable peripheral lung tumor.

DETAILED DESCRIPTION:
The study is aimed to evaluate the efficacy and safety of navigation bronchoscopy guided transbronchial ablation for treating inoperable malignant lung tumor. The study is designed as a single-center prospective trial. The participating centers are Department of pulmonary medicine and endoscopy, Shanghai Chest Hospital,Shanghai Jiao Tong University, China. Patients are divided into two groups, including radiofrequency ablation group and microwave ablation group. Sixty patients are expected to be enrolled into the study with 30 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 year-old.
2. Patients meeting one of the following criteria: 1) patients discovered with peripheral lung lesions that have demonstrated to be lung cancer by pathology with the clinical stage no later than IIA. 2) recurrent or progressive single lesion or solitary intrapulmonary metastasis after surgery, radiotherapy, chemotherapy or other treatment.3) multiple primary lung cancer with the number of tumors no more than 5 and no metastasis. 4) pulmonary metastases with effective treatment of primary disease, the number of metastases no more than 5 and no other metastasis.
3. Chest CT shows the length-diameter of the tumor is more than 8mm and no more than 50mm.
4. Patients are unsuitable for surgery assessed by multidisciplinary team and agree to the primary treatment of ablation.
5. Patients have good compliance and sign the informed consent.

Exclusion Criteria:

1. Patients cannot receive bronchoscopy for the severe cardiopulmonary dysfunction and other indications.
2. Patients have contraindications of general anesthesia.
3. Chest CT or bronchoscopy shows that guided and treatment instruments cannot reach the peripheral lung lesion.
4. There are large blood vessels or important structures adjacent to peripheral lung lesion.
5. Researchers consider the patient do not fit for the study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Local control rate | Three months after ablation
  Local control rate was defined as the proportion of the complete ablation and incomplete ablation of the tumor.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the time of treatment to the time of disease progression or death, assessed up to 1 year
  PFS was defined from the first day after ablation to progression of target lesions and/or appearance of new lesions or death.
Overall survival（OS） | From the time of treatment to the time of the patient death, assessed up to 3 years
  Overall survival（OS) is evaluated after the treatment of ablation until the patient death.
Cancer-specific survival | From the time of treatment to the time of the patient death, assessed up to 3 years
  The cause of death is related to the patient's underlying malignancy.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE 4.0 | From the time of treatment to the complication occured, assessed up to 1 month
  Complications refer to serious operation-related adverse events during and after the operation,such as pneumothorax, bleeding and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris K, Puchalski J, Sterman D. Recent Advances in Bronchoscopic Treatment of Peripheral Lung Cancers. Chest. 2017 Mar;151(3):674-685. doi: 10.1016/j.chest.2016.05.025. Epub 2016 Jun 10. PMID 27292045
- [Background] Koizumi T, Tsushima K, Tanabe T, Agatsuma T, Yokoyama T, Ito M, Kanda S, Kobayashi T, Yasuo M. Bronchoscopy-Guided Cooled Radiofrequency Ablation as a Novel Intervention Therapy for Peripheral Lung Cancer. Respiration. 2015;90(1):47-55. doi: 10.1159/000430825. Epub 2015 May 30. PMID 26044954
- [Background] Jahangeer S, Forde P, Soden D, Hinchion J. Review of current thermal ablation treatment for lung cancer and the potential of electrochemotherapy as a means for treatment of lung tumours. Cancer Treat Rev. 2013 Dec;39(8):862-71. doi: 10.1016/j.ctrv.2013.03.007. Epub 2013 Apr 17. PMID 23601905
- [Background] Wasser EJ, Dupuy DE. Microwave ablation in the treatment of primary lung tumors. Semin Respir Crit Care Med. 2008 Aug;29(4):384-94. doi: 10.1055/s-2008-1081281. PMID 18651356
- [Background] Fernando HC, De Hoyos A, Landreneau RJ, Gilbert S, Gooding WE, Buenaventura PO, Christie NA, Belani C, Luketich JD. Radiofrequency ablation for the treatment of non-small cell lung cancer in marginal surgical candidates. J Thorac Cardiovasc Surg. 2005 Mar;129(3):639-44. doi: 10.1016/j.jtcvs.2004.10.019. PMID 15746749
- [Background] Dupuy DE, Fernando HC, Hillman S, Ng T, Tan AD, Sharma A, Rilling WS, Hong K, Putnam JB. Radiofrequency ablation of stage IA non-small cell lung cancer in medically inoperable patients: Results from the American College of Surgeons Oncology Group Z4033 (Alliance) trial. Cancer. 2015 Oct 1;121(19):3491-8. doi: 10.1002/cncr.29507. Epub 2015 Jun 19. PMID 26096694
- [Background] Ye X, Fan W, Chen JH, Feng WJ, Gu SZ, Han Y, Huang GH, Lei GY, Li XG, Li YL, Li ZJ, Lin ZY, Liu BD, Liu Y, Peng ZM, Wang H, Yang WW, Yang X, Zhai B, Zhang J. Chinese expert consensus workshop report: Guidelines for thermal ablation of primary and metastatic lung tumors. Thorac Cancer. 2015 Jan;6(1):112-21. doi: 10.1111/1759-7714.12152. Epub 2015 Jan 7. PMID 26273346
- [Derived] Xie F, Chen J, Jiang Y, Sun J, Hogarth DK, Herth FJF. Microwave ablation via a flexible catheter for the treatment of nonsurgical peripheral lung cancer: A pilot study. Thorac Cancer. 2022 Apr;13(7):1014-1020. doi: 10.1111/1759-7714.14351. Epub 2022 Feb 14. PMID 35166043